CLINICAL TRIAL: NCT02982577
Title: Effect of Pilocarpine in Patients With Xerostomia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Raony Môlim de Sousa Pereira, MSc, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 27765714.0.0000.5419
Record Dates: First submitted 2016-11-27; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: Xerostomia
Keywords: Xerostomia; Pilocarpine; Quality of life
MeSH Terms: conditions — Xerostomia | interventions — Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilocarpine (Experimental): Spray with Pilocarpine
  Interventions: Drug: Pilocarpine
- Placebo (Placebo Comparator): Spray without Pilocarpine
  Interventions: Other: Spray without Pilocarpine

INTERVENTIONS:
Drug: Pilocarpine — Spray the basis of 1.54% pilocarpine, 3 times per day (each 8 hours), during 90 days.
  Other Names: Pilocarpine spray
  Arms: Pilocarpine
Other: Spray without Pilocarpine — Spray without pilocarpine, 3 times per day (each 8 hours), during 90 days.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a spray the basis of pilocarpine on salivary flow of patients with xerostomia, by radiation therapy, and primary Sjögren's Syndrome treated at the Clinics Hospital of Faculty of Medicine of Ribeirão Preto (HCFMRP-USP), and its impact on quality of life.

DETAILED DESCRIPTION:
There will be two groups: Group 1 (G1) - will use a spray with pilocarpine for three months and after a washout period of a month, use a spray without pilocarpine for another three months; Group 2 (G2) - will use a spray without pilocarpine for three months and after a washout period of a month, use a spray with pilocarpine for another three months (in a randomized, controlled, duble blind and crossover study). Participants will be submitted to OHIP-14, Xerostomia Inventory (XI) and salivary flow measurement before the start of therapy - baseline (T0), one (T2), two (T3) and three (T4) months after starting the use of spray, after washout, crossover occurs and the same parameters are measured for the same periods (T0', T2', T3' and T4'), and is measured one hour after the saliva (T1 and T1') baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or superior to 18 years;
* Both genders;
* Lucid and without diagnosis of any psychiatric disorder;
* Diagnosed with head and neck cancer and treated for a period of up to 5 years with radiotherapy where the major salivary glands (parotid, submandibular and sublingual) were included in the radiation field;
* Primary Sjögren's syndrome with the diagnosis made by the American-European criteria.

Exclusion Criteria:

* Sensitivity to pilocarpine
* Secondary Sjögren's syndrome;
* Type II diabetes mellitus;
* AIDS;
* pregnant or lactating women;
* Glaucoma;
* Uncontrolled asthma;
* Chronic obstructive pulmonary disease;
* Renal diseases;
* Severe cardiovascular diseases;
* Gastrointestinal disorders;
* Hepatic insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Salivary flow | baseline, 1 hour after baseline and each 30 days up to 90 days until start the wash out, and after crossover will repeat these time frame measures
  measured by stimulated salivation

SECONDARY OUTCOMES:
Quality of life | baseline and each 30 days up to 90 days until start the wash out, and after crossover will repeat these time frame measures
  measured by Oral Health Impact Profile (OHIP-14)
Xerostomia grade | baseline and each 30 days up to 90 days until start the wash out, and after crossover will repeat these time frame measures
  measured by Xerostomia Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Camila Tirapelli, PhD, Study Director — University of Sao Paulo
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies AN, Thompson J. Parasympathomimetic drugs for the treatment of salivary gland dysfunction due to radiotherapy. Cochrane Database Syst Rev. 2015 Oct 5;2015(10):CD003782. doi: 10.1002/14651858.CD003782.pub3. PMID 26436597
- [Background] Hanchanale S, Adkinson L, Daniel S, Fleming M, Oxberry SG. Systematic literature review: xerostomia in advanced cancer patients. Support Care Cancer. 2015 Mar;23(3):881-8. doi: 10.1007/s00520-014-2477-8. Epub 2014 Oct 18. PMID 25322971
- [Background] Nikles J, Mitchell GK, Hardy J, Agar M, Senior H, Carmont SA, Schluter PJ, Good P, Vora R, Currow D. Do pilocarpine drops help dry mouth in palliative care patients: a protocol for an aggregated series of n-of-1 trials. BMC Palliat Care. 2013 Oct 31;12(1):39. doi: 10.1186/1472-684X-12-39. PMID 24176001
- [Background] Brito-Zeron P, Siso-Almirall A, Bove A, Kostov BA, Ramos-Casals M. Primary Sjogren syndrome: an update on current pharmacotherapy options and future directions. Expert Opin Pharmacother. 2013 Feb;14(3):279-89. doi: 10.1517/14656566.2013.767333. Epub 2013 Jan 25. PMID 23346917
- [Result] Spivakovsky S, Spivakovsky Y. Parasympathomimetic drugs for dry mouth due to radiotherapy. Evid Based Dent. 2016 Sep;17(3):79. doi: 10.1038/sj.ebd.6401185. PMID 27767109
- [Result] Yang WF, Liao GQ, Hakim SG, Ouyang DQ, Ringash J, Su YX. Is Pilocarpine Effective in Preventing Radiation-Induced Xerostomia? A Systematic Review and Meta-analysis. Int J Radiat Oncol Biol Phys. 2016 Mar 1;94(3):503-11. doi: 10.1016/j.ijrobp.2015.11.012. Epub 2015 Nov 10. PMID 26867879
- [Result] Cheng CQ, Xu H, Liu L, Wang RN, Liu YT, Li J, Zhou XK. Efficacy and safety of pilocarpine for radiation-induced xerostomia in patients with head and neck cancer: A systematic review and meta-analysis. J Am Dent Assoc. 2016 Apr;147(4):236-43. doi: 10.1016/j.adaj.2015.09.014. Epub 2015 Nov 10. PMID 26563850
- [Result] Nikles J, Mitchell GK, Hardy J, Agar M, Senior H, Carmont SA, Schluter PJ, Good P, Vora R, Currow D. Testing pilocarpine drops for dry mouth in advanced cancer using n-of-1 trials: A feasibility study. Palliat Med. 2015 Dec;29(10):967-74. doi: 10.1177/0269216315585473. Epub 2015 May 22. PMID 26001395
- [Result] Wong RK, Deshmukh S, Wyatt G, Sagar S, Singh AK, Sultanem K, Nguyen-Tan PF, Yom SS, Cardinale J, Yao M, Hodson I, Matthiesen CL, Suh J, Thakrar H, Pugh SL, Berk L. Acupuncture-Like Transcutaneous Electrical Nerve Stimulation Versus Pilocarpine in Treating Radiation-Induced Xerostomia: Results of RTOG 0537 Phase 3 Study. Int J Radiat Oncol Biol Phys. 2015 Jun 1;92(2):220-7. doi: 10.1016/j.ijrobp.2015.01.050. Epub 2015 Apr 1. PMID 25841622
- [Result] Tanigawa T, Yamashita J, Sato T, Shinohara A, Shibata R, Ueda H, Sasaki H. Efficacy and safety of pilocarpine mouthwash in elderly patients with xerostomia. Spec Care Dentist. 2015 Jul-Aug;35(4):164-9. doi: 10.1111/scd.12105. Epub 2015 Feb 2. PMID 25639487
- [Result] Noaiseh G, Baker JF, Vivino FB. Comparison of the discontinuation rates and side-effect profiles of pilocarpine and cevimeline for xerostomia in primary Sjogren's syndrome. Clin Exp Rheumatol. 2014 Jul-Aug;32(4):575-7. Epub 2014 Jul 23. PMID 25065774
- [Result] Pimentel MJ, Filho MM, Araujo M, Gomes DQ, DA Costa LJ. Evaluation of radioprotective effect of pilocarpine ingestion on salivary glands. Anticancer Res. 2014 Apr;34(4):1993-9. PMID 24692737
- [Result] Kim JH, Ahn HJ, Choi JH, Jung DW, Kwon JS. Effect of 0.1% pilocarpine mouthwash on xerostomia: double-blind, randomised controlled trial. J Oral Rehabil. 2014 Mar;41(3):226-35. doi: 10.1111/joor.12127. Epub 2013 Dec 30. PMID 24527846